CLINICAL TRIAL: NCT01968408
Title: Effectiveness of Lactobacillus Reuteri DSM 17938 in Preventing Nosocomial Diarrhea in Children: a Randomized, Double-blind Placebo Controlled Trial
Brief Title: Lactobacillus Reuteri DSM 17938 in Preventing Nosocomial Diarrhea in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Hanna Szajewska, Proffesor, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KB/125/2012
Record Dates: First submitted 2012-09-03; First posted 2013-10-24 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Diarrhea
Keywords: nosocomial diarrhea; Lactobacillus reuteri DSM 17938; rotavirus diarrhea; probiotics
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L. reuteri DSM 17938 (Active Comparator): Lactobacillus reuteri DSM 17938,10(9)CFU/daily (for the duration of hospitalization)
  ARM I: Rotavirus vaccinated patients
  ARM II: Non-rotavirus vaccinated patients
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938
- Placebo (Placebo Comparator): Placebo consists of an identical formulation in all respects except that the live probiotic bacteria were excluded
  for the duration of hospitalization
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM 17938 — 10(9) CFU/daily
  Arms: L. reuteri DSM 17938
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
AIM: To determine the efficacy of Lactobacillus reuteri DSM 17938 at a dose of 10(9) CFU for the prevention of nosocomial diarrhea.

TRIAL DESIGN: Double-blind, placebo controlled RCT. INTERVENTION: L reuteri DSM 17938 in a daily dose of 10(9) CFU. PRIMARY OUTCOME: Nosocomial diarrhoea (3 or more loose or watery stools in a 24 h that will occur more than 72 h after admission).

DETAILED DESCRIPTION:
Nosocomial diarrhea is a common problem in hospitalized children. Previously, it has been documented that the administration of L reuteri DSM 17938 at a dose of 10(8) colony forming units (CFU) compared with placebo had no effect on the overall incidence of nosocomial diarrhea (Wanke & Szajewska, J Pediatr 2012). Whether higher doses of L reuteri DSM 17938 have such effects needs to be substantiated in further randomized trials.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-48 mo admitted to the hospital for reasons other than diarrhea
* Signed informed consent.

Exclusion Criteria:

* Acute gastroenteritis within 3 days before admission
* Symptoms other than diarrhea suggesting gastroenteritis
* Use of probiotics within 7 days before admission
* Immunodeficiency disorders
* Breastfeeding >50%
* Underlying gastrointestinal tract disorder
* Malnutrition (weight/high <3pc)

Ages: 1 Month to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2012-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Incidence of nosocomial diarrhea (defined as the passage of 3 or more loose or watery stools in a 24-hour period that will occur more than 72 hours after admission) | Any time starting 72 h after admission

SECONDARY OUTCOMES:
Incidence of diarrhea- passage of 3 or more loose or watery stools in a 24-h period | from the time of admission to the time of discharge of the hospital-expected average 3-5 days
Duration of diarrhea (ie, time till the last loose or watery stool from the onset of diarrhea) | during hospitalisation (expected average 3-5 days) and 72 h after discharge
Need and the length of intravenous rehydration due to diarrhea | During the hospitalization-expected average 3-5 days
Prolongation of the hospitalization due to nosocomial diarrhea | during the hospitalization-expected average 3-5 days
Incidence of rotavirus diarrhea (ie, detection of rotavirus or antigen in the stools) | 72 hours after admission to the hospital to 72 hours after discharge
  Positive test for rotavirus or antigen in the stool sample
Incidence of chronic diarrhea- lasting more than 14 days | untill 14 days after onset of diarrhea
Length of hospital stay | During hospitalisation-expected average 3-5 days
Adverse effects | During hospitalisation (expected average 3-5 days) plus 72 h after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Szajewska, MD, Profesor, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Pediatrics, Medical University of Warsaw, Warsaw, Poland